CLINICAL TRIAL: NCT01183429
Title: 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic Acid for Consolidation of First Remission After Non-Myeloablative Therapy in Patients With High-Risk Neuroblastoma: A Phase II Study
Brief Title: 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic Acid for Consolidation of First Remission After Non-Myeloablative Therapy in Patients With High-Risk Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-159
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-04

CONDITIONS: Neuroblastoma
Keywords: MAB 3F8; RETINOIC ACID (CIS-9 & 13); Bone Marrow; 09-159
MeSH Terms: conditions — Neuroblastoma | interventions — Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3F8 and 13-cis-retinoic acid (Experimental): This phase II, open-label, single arm trial assesses the anti-NB activity of high-dose 3F8 (80 mg/m2/day), which is used in cycles 1-2, with return to standard 3F8 dosage (20 mg/m2/day) in subsequent cycles. Clinical results will be compared to those in the predecessor trials which used only the standard 3F8 dosage. Starting with A(8), patients no longer receive high dose 3F8 but receive only standard dose 3F8 (20mg/m2/day) for all cycles.
  Interventions: Drug: 3F8 and 13-cis-retinoic acid

INTERVENTIONS:
Drug: 3F8 and 13-cis-retinoic acid — 3F8 is dosed at 80 mg/m2/day (cycles 1-2) or 20 mg/m2/day (cycles 3 and beyond) and infused iv over 30-90 minutes. 13-cis-retinoic acid is dosed at 160 mg/m2/day, divided into two doses, x14 days. If a dose is missed, it can be made up at the end of the cycle. It is not taken on same days as 3F8. *High-dose 3F8 will be administered only for patients enrolled on protocol from A(0) to A(7). Starting with A(8), patients receive standard dose (20mg/m2/day) during cycles 1 and 2.

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, the combination of 3F8 and GM-CSF has on the patient and the cancer.

Antibodies are made by the body to attack tumors and to fight infections. 3F8 is the name of one kind of antibody. It is made by mice, and it can attack neuroblastoma in people. 3F8 has been used safely in many patients, and it has killed cancer cells in some patients. One way it can kill cancer cells is by causing the patient's own white blood cells to attack the cancer. Granulocytes are one kind of white blood cell. GM-CSF increases the number of granulocytes in people, and it makes the granulocytes better able to kill the cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NB as defined by a) histopathology (confirmed by the MSKCC Department of Pathology), or b) BM metastases or MIBG-avid lesion(s) plus high urine catecholamine levels.
* High-risk NB as defined by risk-related treatment guidelines1 and the International NB Staging System,89 i.e., stage 4 with (any age) or without (≥18 months of age) MYCN amplification, MYCN-amplified stage 2 or stage 3 (any age), or MYCN-amplified stage 4S.
* The patients are in first CR/VGPR after conventional therapy. They have no measurable MIBG-avid soft tissue tumor assessable for response.
* Signed informed consent indicating awareness of the investigational nature of this program.

Exclusion Criteria:

* Creatinine > 3.0 mg/dL
* ALT, AST and Alkaline Phosphatase > 5.0 times the upper limit of normal
* Bilirubin > 3.0 mg/dL
* Patients with grade 3 or higher toxicities (using the CTCAE v3.0) related to cardiac, neurological, pulmonary or gastrointestinal function as determined by physical exam. Patients must have normal blood pressure for age.
* Progressive disease
* History of allergy to mouse proteins.
* Active life-threatening infection.
* Human anti-mouse antibody (HAMA) titer >1000 Elisa units/ml.
* Inability to comply with protocol requirements

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-08-12 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2018-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kushner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Kushner BH, Modak S, Basu EM, Roberts SS, Kramer K, Cheung NK. Posterior reversible encephalopathy syndrome in neuroblastoma patients receiving anti-GD2 3F8 monoclonal antibody. Cancer. 2013 Aug 1;119(15):2789-95. doi: 10.1002/cncr.28137. Epub 2013 Apr 30. PMID 23633099
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3F8 and 13-cis-retinoic Acid
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 3F8 and 13-cis-retinoic Acid
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33
  Colombia | 1
  Greece | 1
  India | 1
  Singapore | 1
  Spain | 2

OUTCOME MEASURES:

1. Primary Outcome: Assess the Impact of High-dose 3F8/GM-CSF
Description: on relapse-free survival in patients in first complete or very good partial remission, but at high risk of relapse.
Time Frame: 2 years
Population: No data were collected
Arm/Group | 3F8 and 13-cis-retinoic Acid
Number analyzed (Participants) | 0

2. Secondary Outcome: Apply Real-time Quantitative RT-PCR
Description: to test the hypothesis that the minimal residual disease content of bone marrow after the first treatments with 3F8/GMCSF has significant prognostic impact on relapse-free survival.
Time Frame: 2 years
Population: No data were collected
Arm/Group | 3F8 and 13-cis-retinoic Acid
Number analyzed (Participants) | 0

3. Secondary Outcome: Monitor Safety of the High-dose Antibody Treatment
Description: to assure no side-effects or noxious sequelae develop or emerge that were not seen in the prior phase I study.
Time Frame: 2 years
Population: No data were collected
Arm/Group | 3F8 and 13-cis-retinoic Acid
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: N/A Data were not collected
Description: Data were not collected
Arm/Group | 3F8 and 13-cis-retinoic Acid
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-24): https://cdn.clinicaltrials.gov/large-docs/29/NCT01183429/Prot_SAP_000.pdf